CLINICAL TRIAL: NCT02145923
Title: Effectiveness and Safety of Intravenous Infusion of Bone Marrow Derived Allogeneic Multipotent Mesenchymal Stromal Cells for Enhancing Hematopoietic Recovery and Prophylaxis of Neutropenic Enterocolitis in Hematological Patients With Aplasia After High-dose Chemotherapy.
Brief Title: Effectiveness and Safety of MMSCs for Enhancing Hematopoietic Recovery and Prophylaxis of Neutropenic Enterocolitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Principal Investigator, Zarui Simavonyan, MD, Burnasyan Federal Medical Biophysical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RU-FMBC-05-01-14
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Neutropenic Enterocolitis; Myeloablative Chemotherapy Induced Bone Marrow Aplasia
Keywords: Hodgkin Lymphoma; Non-Hodgkin's Lymphomas; Allogeneic Mesenchymal Stem Cell Transplantation; Autologous Peripheral Blood Stem Cell Transplantation; Neutropenic Enterocolitis; Myeloablative Chemotherapy; Bone Marrow Aplasia
MeSH Terms: conditions — Enterocolitis, Neutropenic; Hodgkin Disease; Anemia, Aplastic | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- allogeneic MMSCs infusion (Other): Subjects will undergo peripheral blood stem cell mobilisation and collection with subsequent high-dose chemotherapy. After finalization of high-dose chemotherapy subjects will receive bone marrow derived allogeneic multipotent mesenchymal stromal cells intravenous infusion two hours prior to autologous peripheral blood cells infusion.
  Interventions: Procedure: Peripheral blood stem cell mobilisation and collection; Drug: High-dose chemotherapy; Drug: Bone marrow derived allogeneic MMSCs infusion; Procedure: Autologous peripheral blood stem cells infusion

INTERVENTIONS:
Procedure: Peripheral blood stem cell mobilisation and collection
Drug: High-dose chemotherapy — High-dose chemotherapy will be performed according to protocols ICE and BEAM (standard scheme)
Drug: Bone marrow derived allogeneic MMSCs infusion
Procedure: Autologous peripheral blood stem cells infusion

SUMMARY:
Subjects will undergo peripheral blood stem cell mobilisation and collection with subsequent high-dose chemotherapy. After finalization of high-dose chemotherapy subjects will receive bone marrow derived allogeneic multipotent mesenchymal stromal cells intravenous infusion two hours prior to autologous peripheral blood cells infusion. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Patients with verified diagnosis Hodgkin's lymphoma or non-Hodgkin's lymphoma will undergo peripheral blood stem cell mobilisation and collection (chemotherapy + G-CSF or G-CSF+Plerixafor).

After that high-dose chemotherapy will be performed according to protocols ICE and BEAM (standard scheme).

Patient will receive bone marrow derived allogeneic multipotent mesenchymal stromal cells infusion 48 hours after last administration of cytotoxic agent . Number of cells calculated according to patient's body weight (1,5-2,0 mln of cells/kg), time of infusion - 30 minutes. Two hours later patient will receive autologous peripheral blood cells infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from Hodgkin's lymphoma, non-Hodgkin's lymphoma with complete or partial remission.
* Patient is candidate to high-dose chemotherapy with subsequent autologous hematopoietic stem cell transplantation.
* Absence of infection, cardiovascular, respiratory, renal and hepatic dysfunctions, focal neurological symptoms.
* Karnofsky score at least 70.
* Patient successfully undergone mobilization of peripheral blood stem cells.
* Patient is familiar with Participant information sheet.
* Patient signed informed consent form.

Non-inclusion Criteria:

* Severe chronic comorbidity with symptoms of organ or system failure.
* Significant abnormalities in laboratory tests.
* Participation in other clinical trials (or intake of study drugs) within prior 3 months.
* Conditions restricting commitment to participating in the trial (dementia, neuropsychiatric disorders, drug and alcohol abuse)
* Patients with malignant solid tumors.
* Patients with medical history of heterotopic ossification.

Exclusion Criteria:

* Progression or relapse of lymphoma during therapy.
* Confirmed syphilis, HIV, hepatitis B or C infection
* Absence of clinical and laboratory signs of hematopoietic recovery and persistent enterocolitis at day 14 after the manipulation (Visit 15). While the patient remains in the hospital and continues treatment according to requirements of standard therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events (SAEs) and serious adverse reactions (SARs) | 2 weeks after treatment

SECONDARY OUTCOMES:
Time of hematopoietic recovery | Follow up to completion (up to 3 months after treatment)
  Monitoring of time of hematopoietic recovery assessed by complete blood count
Neutropenic enterocolitis | Follow up to completion (up to 3 months after treatment)
  Monitoring of frequency (number of participants) and severity of neutropenic enterocolitis during the study period
Infectious complications | Follow up to completion (up to 3 months after treatment)
  Monitoring of frequency and severity of infectious complications during the study period. Frequency of infectious complications will be represented in number of infections verified by clinical, instrumental examination and/or laboratory methods.
Transfusion needs | Follow up to completion (up to 3 weeks after treatment)
  Monitoring of frequency (number of participants) of transfusion needs during neutropenic period

CONTACTS AND LOCATIONS:
Overall Officials: Zaryi Simavonyan, MD, Principal Investigator — Burnasyan Federal Medical Biophysical Center; Ilya I Eremin, MD, PhD, Principal Investigator — Burnasyan Federal Medical Biophysical Center
Locations (1):
- State Research Center Burnasyan Federal Medical Biophysical Center FMBA of Russia, Moscow, Russia